CLINICAL TRIAL: NCT02788656
Title: PARENT Trial Pilot Pulmonary Artery Pressure Reduction With ENTresto (Sacubitril/Valsartan)
Brief Title: Pulmonary Artery Pressure Reduction With ENTresto (Sacubitril/Valsartan)
Acronym: PARENT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate Recruitment
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Akshay Desai, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P000831/MGH
Record Dates: First submitted 2016-05-23; First posted 2016-06-02 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Congestive Heart Failure
Keywords: heart failure; neprilysin; implantable hemodynamic monitor; angiotensin-receptor blocker; angiotensin-converting enzyme inhibitor
MeSH Terms: conditions — Heart Failure | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin II Type 1 Receptor Blockers; Angiotensin Receptor Antagonists; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Group A will receive sacubitril/valsartan + placebo for weeks 1-12. and then sacubitril/valsartan only for weeks 13-32. All subjects in Group A will also receive longitudinal pulmonary artery pressure monitoring using a previously placed implantable hemodynamic monitor (CardioMEMS device).
  Interventions: Device: Implantable Hemodynamic Monitor; Drug: sacubitril/valsartan
- Group B (Active Comparator): Group B will receive an Angiotensin-Converting Enzyme Inhibitor (ACEi) or Angiotensin II Type 1 Receptor Blocker (ARB) + placebo for weeks 1-6 (depending on previous background therapy) and then switch to sacubitril/valsartan + placebo for weeks 7-12.
  Group B will then receive sacubitril/valsartan only for weeks 13-32. All subjects in Group B will also receive longitudinal pulmonary artery pressure monitoring using a previously placed implantable hemodynamic monitor (CardioMEMS device).
  Interventions: Device: Implantable Hemodynamic Monitor; Drug: Angiotensin-Converting Enzyme Inhibitor; Drug: Angiotensin II Type 1 Receptor Blocker; Drug: sacubitril/valsartan

INTERVENTIONS:
Device: Implantable Hemodynamic Monitor — The CardioMEMS device is an implantable pulmonary artery pressure monitor that is FDA-approved for use in patients with symptomatic heart failure and previous heart failure hospitalization. Patients eligible for this study are those with an already implanted CardioMEMS device.
  Other Names: CardioMEMS
Drug: Angiotensin-Converting Enzyme Inhibitor — Conventional, guideline-directed therapy for heart failure and reduced ejection fraction
  Other Names: ACE inhibitor, ACEi
  Arms: Group B
Drug: Angiotensin II Type 1 Receptor Blocker — Conventional, guideline-directed therapy for heart failure and reduced ejection fraction in ACE-inhibitor intolerant patients
  Other Names: Angiotensin Receptor Blocker, ARB
  Arms: Group B
Drug: sacubitril/valsartan — Angiotensin-neprilysin inhibitor that is now FDA-approved and guideline-directed therapy for patients with symptomatic heart failure and reduced ejection fraction despite treatment with an ACE-inhibitor/Angiotensin-Receptor Blocker
  Other Names: Entresto

SUMMARY:
This pilot study will assess the impact of sacubitril/valsartan (trade name Entresto) on the elevated pulmonary artery pressures in patients with heart failure with reduced ejection fraction, measured using a previously implanted hemodynamic monitoring device (CardioMEMS).

DETAILED DESCRIPTION:
Angiotensin-converting enzyme inhibitors (ACEi) have been a cornerstone treatment for patients with heart failure and reduced ejection fraction (HFrEF) for over 25 years. They are included in every major set of guidelines for HFrEF management. Angiotensin receptor blockers (ARB's, such as valsartan) have similarly been shown to decrease the mortality rate of patients with HFrEF for patients who are unable to tolerate ACEi therapy.

The newest neurohormonal therapy approved for heart failure (August 2015) is sacubitril/valsartan (trade name Entresto). This medication is the first of a new family of agents (ARNI = angiotensin receptor antagonist with neprilysin inhibitor), combining the approved angiotensin receptor blocker valsartan with sacubitril, an inhibitor of neprilysin, which is a neutral endopeptidase that degrades endogenous vasoactive peptides. Treatment with sacubitril increases circulating levels of natriuretic peptides, which have been shown to facilitate natriuresis and vasodilation. Although the precise mechanisms responsible for benefit in heart failure remain unclear, sacubitril/valsartan may reduce the fluid retention and vasoconstriction that contribute to heart failure symptoms, and may also decrease apoptosis and remodeling that lead to disease progression. There is limited data about the incremental acute and long-term hemodynamic effects of composite neprilysin/angiotensin-receptor inhibitors over enalapril, and these data may provide important mechanistic insights.

Progress in HF management outside the hospital has included validation of a strategy of ongoing monitoring of pulmonary artery pressures every day from home via a monitor implanted in a distal pulmonary artery, the CardioMEMS device. The information is transmitted to a website where it is reviewed by the HF team, who can intervene to adjust diuretics and other medications by phone to avert decompensation and re-hospitalization. The device received FDA approval in mid 2014, and is now being implanted in many cardiac catheterization laboratories, including at Brigham and Women's Hospital. The pressure information is reviewed regularly by the HF management team who are in regular contact with the patient to aid in management decisions.

In summary, this pilot study will assess the impact of sacubitril/valsartan, an approved drug for heart failure with reduced ejection fraction (HFrEF) on the elevated pulmonary artery pressures measured using an implanted monitoring device that is also approved for such patients. Both the medication and the device will be used according to approved indications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to provide written informed consent
2. Patients ≥18 years of age, male or female, in NYHA Class II- III HF, previously hospitalized for HFrEF with LVEF < 35% (measured within the past year), and who have no subsequent LVEF>35%.
3. Systolic BP > 95 mm Hg at most recent clinical assessment.
4. Stable, ambulatory patients without the need for change in diuretics and other HF drugs (RAS blockers, beta blockers or mineralocorticoid receptor blockers) during the past 5 days
5. CardioMEMS HF System implanted for NYHA Class III HF. Patient transmitting information regularly and system functioning appropriately.
6. NT-proBNP > 500 pg/ml within 90 days of CardioMEMS implantation.
7. Average PAPm >20mm Hg during the 7 days prior to enrollment, including at least 4 daily measurements.
8. Women of childbearing age must be on highly effective method of contraception

Exclusion Criteria:

1. Treatment with vasodilators (other than nitrates, hydralazine) and/or IV inotropic drugs.
2. Entresto taken within the past 30 days.
3. History of hypersensitivity, intolerance or angioedema to previous renin-angiotensin system (RAS) blocker, ACE inhibitor, ARB, or Entresto.
4. eGFR < 30 ml/min/1.73 m2 as measured by the simplified MDRD formula.
5. Serum potassium > 5.5 mmol/L.
6. Acute coronary syndrome, stroke, transient ischemic attack, cardiovascular surgery, PCI, or carotid angioplasty within the preceding 3 months.
7. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within 3 months after trial entry.
8. Non-cardiac condition(s) as the primary cause of dyspnea.
9. Implantation of a cardiac resynchronization therapy device (CRT/D) within the pr preceding 3 months or intent to implant a CRT/D, which may alter the pressures during the course of the study.
10. History of heart transplantation, placement of an LVAD, listing for Status IA for cardiac transplantation or planned placement of an LVAD within 3 months following randomization.
11. Documented untreated ventricular arrhythmia with syncopal episodes within the prior 3 months.
12. Symptomatic bradycardia or second or third degree heart block without a pacemaker.
13. Hepatic dysfunction, as evidenced by total bilirubin > 3 mg/dl.
14. Pregnancy
15. Women who are breastfeeding
16. Chronic lithium use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren G Gilstrap, MD, Study Director — Brigham & Womens' Hospital
Locations (1):
- Brigham and Women's Hospita, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Entresto + Placebo
- Group B: ACE/ARB + Placebo
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [45 to 70] | 66.5 [63 to 70] | 62 [45 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
mean PA Pressure [Mean (Full Range); unit: mm Hg] | 24 [21 to 27] | 28 [20 to 36] | 26 [20 to 36]
NTproBNP [Mean (Full Range); unit: pg/mL] | 634 [235 to 1032] | 750 [202 to 1297] | 692 [202 to 1297]

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Mean Change in Mean Pulmonary Artery Pressure (PAPm) With Sacubitril/Valsartan Compared to the Mean Change in PAPm With Continued ACEi/ARB
Description: Change in mean PAP in group A versus group B
Time Frame: Baseline, 6 weeks
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 2
mm Hg | 0 [0 to 0] | -2.5 [-11 to 6]

2. Primary Outcome: The Acute Change in PAPm After the First Administration of Sacubitril/Valsartan
Description: Change in PAPm at 3 hours
Time Frame: Baseline, 3 hours (after first dose of sacubitril/valsartan)
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 2
mm Hg | -3.5 [-8 to 1] | -15 [-15 to -15]

3. Secondary Outcome: Mean Change in PAPm in Both Groups on Sacubitril/Valsartan
Description: Change in PAPm from week 12-32
Time Frame: 20 weeks (weeks 12 to 32 of the study)
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 1 | 2
mm Hg | 6 [6 to 6] | 2 [1 to 3]

4. Secondary Outcome: The Difference Between Mean Change in PAPm From Baseline on Sacubitril/Valsartan Compared to ACEI/ARB
Description: Change in PAPm on sacubitril/valsartan: Measured from baseline to week 6 (group A) and week 7-week 12 (Group B)
Time Frame: 6 weeks (week 1-6 of the study for group A, weeks 7-12 for group B)
Measure: Mean (Full Range); unit: mm Hg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 2
mm Hg | 0 [0 to 0] | 1.5 [0 to 3]

5. Secondary Outcome: Determine the Change in Distance Walked During a Standard 6 Minute Walk Test From Baseline
Description: Change in 6 minute walk distance in Group A vs. Group B at 6 weeks
Time Frame: Baseline, 6 weeks
Measure: Mean (Full Range); unit: m
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 2
m | 36 [8 to 63] | -5 [-30 to 20]

6. Secondary Outcome: Change in NT-proBNP
Description: Change in NT-proBNP from baseline to 6 weeks
Time Frame: Baseline
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 2
pg/mL | -85 [-136 to -33] | 250 [-15 to 515]

7. Other Pre Specified Outcome: The Relationship of Change in PAPm to Change in the Questions in the Kansas City Cardiomypathy Questionnaire (KCCQ) 3,7,8,9
Description: Correlation between change in PAPm and change in KCCQ at 32 weeks
Time Frame: Baseline, 32 weeks (testing performed at intervals during study)
Population: Not reported due to lack of adequate data (too few participants enrolled)
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Mean Change in Total Daily Diuretic Dose While on Sacubitril/Valsartan
Description: Mean change in total daily diuretic dose while on sacubitril/valsartan (32 weeks)
Time Frame: Baseline, 32 weeks (testing performed at intervals during study)
Population: ** Data not reported as too few participants were enrolled for meaningful analysis (n=4)
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: No difference from standard definitions
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=2) | Group B (N=2)
Heart Failure Hospitalization (Cardiac disorders) | 1 (1) | 0 (0) — Hospitalization for worsening heart failure

LIMITATIONS AND CAVEATS:
Study terminated after enrollment of 4 patients due to lack of enrollment. Limited number of participants limits meaningful generalization of study results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT02788656/Prot_SAP_000.pdf